CLINICAL TRIAL: NCT02618993
Title: Effects of the Bilateral Mandibular Nerve Block (V3) in Mandibular Osteotomy: a Prospective, Randomized, Double-blind Versus Placebo Study
Brief Title: Effects of the Bilateral Mandibular Nerve Block (V3) in Mandibular Osteotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9560; 2015-001345-88 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-12-02 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Mandibular Fracture Trauma; Orthognathic Surgery; Maxillofacial Osteotomy
Keywords: mandibular nerve block; mandibular osteotomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Control group: Realization of the V3 block with a placebo in maxillofacial surgeries
  Interventions: Procedure: Realization of the V3 block in maxillofacial surgeries
- Loco-regional anesthesia (LRA) group (Experimental): Loco-regional anesthesia (LRA) group: Realization of the V3 block with Ropivacaine in maxillofacial surgeries
  Interventions: Procedure: Realization of the V3 block in maxillofacial surgeries

INTERVENTIONS:
Procedure: Realization of the V3 block in maxillofacial surgeries — bilateral mandibular block in maxillofacial surgeries

SUMMARY:
The sensory innervation of the face depends on the trigeminal (fifth cranial) which is divided into three branches, the mandibular nerve (V3) having motor fibers to the temporal and masseter muscle. The regional anesthesia of the face has grown in recent years for performing certain actions under light general anesthesia or sedation. The mandibular block is a simple and reliable technique but little used. Yet it reduces postoperative pain sagittal osteotomy of the mandibular branch by reducing consumption of opioids and in the oropharynx cancer surgery. Made with ropivacaine, known for its vasoconstrictive action, it also improves the visibility of the operative field during mandibular osteotomies reducing bleeding. Despite a real clinical benefit (ease of implementation, latency and duration of action of the local anesthetic), the V3 block ropivacaine is not evaluated in the maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients and patients from 15 to 18 years old
* with mandibular trauma or orthognathic surgery
* Affiliated to a national insurance scheme
* to have signed the informed consent of this study
* Physical status score 1-3

Exclusion Criteria:

* allergy to local anesthetics
* severe coagulopathy
* hypovolemic patient
* Protected minor or major patients or in the incapacity to give his consent according to the article L1121-8 of the Code of the Health Public.
* Pregnant or breast-feeding women according to the article L1121-5 of the Code of the Health Public.
* Vulnerable People.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
consumption of morphine (cumulative dose) during the first post operative 24 hours valued in mg | 1 day
consumption of morphine (cumulative dose) during the first post operative 24 hours detected thanks to the "Patient Controlled Analgesia" | 1 day

SECONDARY OUTCOMES:
Tolerability : effects of the block on nausea / vomiting (consumption of antiemetic in mg) during the first post operative 24 hours | 1 day
Postoperative pain valued thanks to Visual Analog Scale (VAS), VAS max in post anesthesia care units (PACU) every 30 minutes and in department every 4 hours | 1 day
postoperative bleeding (in mL) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François PERRIGAULT, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Hôpital Gui de Chauliac, Montpellier, France

REFERENCES:
- [Derived] Bertuit M, Rapido F, Ly H, Vannucci C, Ridolfo J, Molinari N, De Boutray M, Galmiche S, Dadure C, Perrigault PF, Capdevila X, Chanques G. Bilateral mandibular block improves pain relief and morphine consumption in mandibular osteotomies: a prospective, randomized, double-blind, placebo-controlled clinical trial. Reg Anesth Pain Med. 2021 Apr;46(4):322-327. doi: 10.1136/rapm-2020-102417. Epub 2021 Feb 9. PMID 33563767